CLINICAL TRIAL: NCT00247117
Title: Study of the Effect of Metformin in Patients With Non-Alcoholic Fatty Liver Disease
Brief Title: Metformin in Patients With Non-Alcoholic Fatty Liver Disease (NAFLD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaplan Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 037-2003
Record Dates: First submitted 2005-10-31; First posted 2005-11-01 (Estimated); Last update posted 2006-10-09 (Estimated); Status verified 2003-10

CONDITIONS: Liver Diseases
Keywords: non-alcoholic fatty liver disease; insulin resistance; metformin
MeSH Terms: conditions — Liver Diseases; Non-alcoholic Fatty Liver Disease; Insulin Resistance | interventions — Metformin

INTERVENTIONS:
Drug: Metformin

SUMMARY:
The purpose of this study is to examine the effect of metformin on biochemical and histological findings in NAFLD patients with insulin resistance syndrome.

DETAILED DESCRIPTION:
Study population:

30 patients will be included who meet all the following criteria: ALT > 2 times normal range; liver histology revealing NASH (type 2-4), without cirrhosis; clinical characteristics of the metabolic syndrome as defined by the NCEP, but no overt diabetes; negative work-up for other causes of liver diseases including alcohol intake < 40 g/week.

All patients will undergo liver biopsy and only patients with type 2-4 (steatosis + inflammation, or steatosis plus ballooning degeneration, or steatosis plus fibrosis and/or Mallory bodies) but without cirrhosis will be included.

Patients who received lipid lowering medications or anti hypertensive drugs prior to study will continue the treatment. Patients who will develop overt type 2 DM with HbAic > 7% during study will be withdrawn.

Intervention:

All patients will have dietary intervention by a dietician and will be encouraged to increase physical activity. Patients will be receiving metformin 850 mg tid for 12 months.

Outcome:

* Improvement of liver enzymes (ALT, AST, GGT)
* Improvement of metabolic profile: lipid profile, fasting and post-load glucose and insulin levels, HOMA.
* Liver histology (repeated liver biopsy after 1 year).
* Soluble TNF receptors- TNF-receptor P55 and P75.

ELIGIBILITY:
Inclusion Criteria:

* ALT > 2 times normal range.
* Liver histology revealing non-alcoholic steatohepatitis [NASH] (type 2-4), without cirrhosis.
* Clinical characteristics of the metabolic syndrome as defined by the National Cholesterol Education Program (NCEP), but no overt diabetes.
* Negative work-up for other causes of liver diseases including alcohol intake < 40 g/week.

Exclusion Criteria:

* Diabetes mellitus.
* Alcohol intake > 40 g per week.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15
Dates: Start 2004-01; Study Completion 2005-08

PRIMARY OUTCOMES:
histological and biochemical changes

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Malnick, MD, Study Director — Kaplan Medical Center
Locations (1):
- Institute of Endocrinology, Kaplan Medical Center, Rehovot, Israel